CLINICAL TRIAL: NCT07132190
Title: A Double-Blind Phase II Randomized Study of Adaptively Delivered LINAC-Based Stereotactic Radiation for Volatile Brain Metastases With Same-Day Planning and Margin Reduction
Brief Title: Stereotactic Radiation for Growing/Changing Brain Metastases With Same-Day Radiation Planning and Treatment With Margin Reduction
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ayal A. Aizer, MD (Other)
Collaborators: Varian, a Siemens Healthineers Company (Industry)
Responsible Party: Sponsor-Investigator, Ayal A. Aizer, MD, Director, Central Nervous System Radiation Oncology; Associate Professor, Harvard Medical School, Brigham and Women's Hospital
Organization: Brigham and Women's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 25-133
Record Dates: First submitted 2025-08-04; First posted 2025-08-20 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Brain Metastases, Adult; Brain Tumor - Metastatic; Brain Metastases From Non-small Cell Lung Cancer (NSCLC); Brain Metastases From Extra-cranial Solid Tumors
Keywords: Brain Mets; Brain Metastases; Brain-directed stereotactic radiation; Brain radiation; Volatile Brain Metastases; Intracranial lesion; SRS; SRT; RANO; PTV; Planning Target Volume; Local Recurrence; Radiation Necrosis; Adaptive; VMAT; Volumetric Modulated Arc Therapy; Margin; Volatile; Rapid; Growth; Shift; neurocognitive; quality of life; survival; same day; randomized
MeSH Terms: conditions — Brain Neoplasms; Margins of Excision; Fasting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- 0mm PTV (Experimental): 0mm uncertainty margin
  Interventions: Radiation: Linear accelerator-based stereotactic radiation for brain metastases using 0mm or 1mm PTV
- 1mm PTV (Active Comparator): 1mm uncertainty margin
  Interventions: Radiation: Linear accelerator-based stereotactic radiation for brain metastases using 0mm or 1mm PTV

INTERVENTIONS:
Radiation: Linear accelerator-based stereotactic radiation for brain metastases using 0mm or 1mm PTV — Linear accelerator-based stereotactic radiation for brain metastases using 0mm or 1mm PTV
  Other Names: SRS; SRT

SUMMARY:
The goal of this study is to evaluate the feasibility and effectiveness of same-day radiation planning and treatment. The study will shorten the time interval between radiation planning (radiation mapping) and radiation treatment. The intent of this shorter time interval is to increase the likelihood that the brain metastases being treated remain fully within the high-dose radiation fields.

Participants will be randomized to receive brain-directed stereotactic radiation with a 1mm margin or 0mm margin, have their simulation/radiation planning imaging on the same day that brain-directed stereotactic radiation is delivered, and have repeat simulation/radiation planning scans during the course of treatment if more than 2-3 days have elapsed since the most recent scans.

DETAILED DESCRIPTION:
Adaptively designed radiation, which adjusts a given radiation plan for real time changes in patient position or anatomy, has become a standard approach within many oncologic entities to combat the effect of shifts between simulation and treatment. Adaptively planned SRS/SRT with same day brain MRI and treatment delivery offers potential to quantify the impact of treatment planning time while also reducing margins and potentially improving rates of local recurrence and radiation necrosis. This trial aims to explore the viability of adaptively designed SRS/SRT with same day planning and treatment in combination with tighter planning margins in both controlling brain metastases locally and minimizing the risk of radiation necrosis in a phase 2 randomized study.

Participants will have a preliminary stereotactic treatment plan created from a diagnostic brain MRI indicating the need for treatment. The preliminary plan will undergo departmental-standard physics, therapy, and quality assurance checks, spanning a total of 1-2 weeks, after which the patient will return for treatment. On the day of treatment (SRS) or start of treatment (SRT), a repeat MRI brain will be performed for planning purposes on an MRI simulator. A synthetic computed tomography (CT) scan will be generated from the new MRI. The previously generated contours and plan will be adapted to the new MRI and the fused synthetic CT. Lastly, the treatment will be delivered.

The primary objective is to assess the percentage of patients that demonstrate tumor beyond the standard planning margin (1.0mm PTV) at the time of stereotactic treatment.

An important secondary objective is to quantify local recurrence and radiation necrosis rates in patients treated with same day simulation and treatment, based on randomization to a PTV of 0mm or 1.0mm.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have a biopsy proven solid malignancy with at least one intact, residual or recurrent, intracranial lesion radiographically consistent with or pathologically proven to be a brain metastasis meeting one of the following criteria:

   1. Growth of 1.0mm per week or more, on average, based on the two most recent brain MRIs preceding study enrollment
   2. Abutment, to within 1.0cm, of a region of intracranial edema
   3. Proximity (within 5.0cm) to a surgical cavity created within 30 days of enrollment
   4. Proximity (within 5.0cm) to another source of physical displacement
2. Age of at least 18 years
3. Karnofsky performance status of at least 60
4. Estimated survival of at least 3-6 months in the opinion of the enrolling clinician and/or study PI
5. Ability to understand and the willingness to sign a written informed consent document by either ink on paper or a DF/HCC approved eConsent medium

Exclusion Criteria:

1. Participants who cannot tolerate a brain MRI
2. Patients who cannot receive gadolinium
3. Participants with end stage renal disease
4. Participants with widespread, definitive leptomeningeal disease
5. Pregnant women are excluded from this study because of the potential deleterious effects of gadolinium on the developing fetus. Because there is an unknown but potential risk for adverse events in nursing infants, women who are breastfeeding are not eligible for this study as well

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
To assess the percentage of patients that demonstrate tumor beyond the standard planning margin (1.0mm PTV) at the time of stereotactic treatment. | Diagnostic MRI to MRI on first day of treatment
  Percentage of patients, based on clinical and radiographic assessment, in which the repeat same day/simulation MRI reveals tumor extending beyond a 1.0mm PTV margin of the plan developed on the diagnostic MRI (i.e. the percentage of patients for which the MRI obtained on the same or first day of treatment displays tumor extending 1.0mm beyond the extent of the tumor on the planning MRI).

SECONDARY OUTCOMES:
Overall survival | Duration of time on study (estimated 1 year)
  Clinical parameter
Death due to neurologic disease progression | Duration of time on study (estimated 1 year)
  Clinical assessment via review of study visits and medical records indicating cause of death (neurologic versus non-neurologic)
Performance status | Duration of time on study (estimated 1 year)
  Karnofsky performance status (KPS), assessed longitudinally. A higher score indicates better functional status and less dependence on others.
Progression free survival | Duration of time on study (estimated 1 year)
  Clinical assessment of first progression after treatment
Quality of life/symptom burden and interference | Duration of time on study (estimated 1 year)
  Questionnaire - MD Anderson Symptom Inventory - Brain Tumor (MDASI-BT). Assessed longitudinally.
  Scored by calculating the mean of the 13 core symptom items and the mean of the 6 interference items. A 0-10 scoring scale is used, with 0 representing an item is not present and 10 representing the highest severity. An item rated 5 or higher may indicate a moderate-to-severe symptom or interference.
Neurocognitive function via Hopkins Verbal Learning Test-Revised | Baseline to 12 months after baseline
  Hopkins Verbal Learning Test-Revised (HVLT-R) scored by number of words recalled. Larger number represents better neurocognitive function. T and Z scores derived using number of words recalled
Time to detection of new brain metastases | Duration of time on study (estimated 1 year)
  Time from treatment to first appearance of new brain metastases on radiographic assessment
Time to development of radiation necrosis | Duration of time on study (estimated 1 year)
  Time from treatment to first appearance of new necrosis on radiographic assessment
Time to development of leptomeningeal disease | Duration of time on study (estimated 1 year)
  Time from treatment to first appearance of leptomeningeal disease on radiographic assessment
Time to local recurrence | Duration of time on study (estimated 1 year)
  Time from treatment to first appearance of local recurrence on radiographic assessment
Time to salvage craniotomy | Duration of time on study (estimated 1 year)
  Time from treatment to first use of craniotomy as salvage therapy
Time to additional radiotherapeutic treatments after the initial course | Duration of time on study (estimated 1 year)
  Time from treatment to first use of additional radiotherapeutic treatments after the initial course
Time to the development of seizures | Duration of time on study (estimated 1 year)
  Time from treatment to development of primary seizures on clinical assessment
Neurocognitive function via Trail Making Test Part A and B (TMT) | Baseline to 12 months after baseline
  Trail Making Test Part A and B (TMT) scored based on time to completion of assessment. Shorter time interval reflects better neurocognitive function
Neurocognitive function via Controlled Word Association Test (COWAT) | Baseline to 12 months after baseline
  Controlled Word Association Test (COWAT) scored by number of words patient can produce in one minute. Larger number of words represents better neurocognitive function
Neurocogntive function via Mini Mental Status Examination (MMSE) | Baseline to 12 months after baseline
  Mini Mental Status Examination (MMSE) scored by sum of components within assessment. Higher score represents better neurocognitive function.

CONTACTS AND LOCATIONS:
Overall Officials: Ayal A Aizer, MD, MHS, Principal Investigator — Dana-Farber/Brigham and Women's Cancer Center
Locations (1):
- Brigham and Women's Hospital / Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided